CLINICAL TRIAL: NCT00686114
Title: Concurrent Chemoradiotherapy Containing Paclitaxel and Cisplatin With/Without Tarceva in Locally Advanced Esophageal Carcinoma: a Randomized Phase III Multi-center Trial.
Brief Title: Concurrent Chemoradiotherapy Containing Paclitaxel&Cisplatin With/Without Tarceva in Locally Advanced Esophageal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Wu Shixiu, Professor, Wenzhou Medical University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Shixiu - 1
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; chemoradiation; radiosensitivity; EGFR inhibition
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel; Cisplatin; Erlotinib Hydrochloride; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental): Enlarged field + Paclitaxel + Cisplatin + Tarceva
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Drug: Tarceva; Radiation: Radiotherapy
- B (Experimental): Enlarged field + Paclitaxel + Cisplatin
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Radiation: Radiotherapy
- C (Active Comparator): Conventional field + Paclitaxel + Cisplatin + Tarceva
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Drug: Tarceva; Radiation: Radiotherapy
- D (Active Comparator): Conventional field + Paclitaxel + Cisplatin
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Paclitaxel — 135mg/m2, day 1 and day 29 of the radiotherapy.
Drug: Cisplatin — 20mg/m2, days 1-3,days 29-31 from the beginning of radiotherapy.
Drug: Tarceva — 150mg/day,oral administration, from day 1 to day 42 (at the beginning of therapy)
  Other Names: Erlotinib Hydrochloride Tablets
  Arms: A; C
Radiation: Radiotherapy — Enlarged field radiotherapy
  Arms: A; B
Radiation: Radiotherapy — Conventional field radiotherapy
  Arms: C; D

SUMMARY:
This study is multi-center randomized phase III one to evaluate the difference in local-control and survival rate between patients receiving concurrent chemoradiotherapy combined Tarceva or not.

DETAILED DESCRIPTION:
For the esophageal carcinoma in II~III stage, routine dosage of Paclitaxel and platinum medicine chemotherapy concurrently radical radiotherapy is worthy to be studied. On this base, we advanced approach the enlarged field radiotherapy and the intervention of Tarceva. And we approach the therapeutic effect for this method theoretically, which may give a further reasonable guidance for the clinical therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be confirmed Esophageal Carcinoma pathologically
2. (EUS)I～IVa, without contraindication for radical radiotherapy
3. Subjects haven't been given neither radiotherapy nor chemotherapy before
4. Age 18-70,behavioral status evaluation ECOG scores 0-2 and anticipated survival more than 6 months
5. In 7 days after being selected, subjects should follow the status: WBC ≥ 4.0 x 10^9/L; ANC ≥ 1.5x 10^9/L; PLT ≥ 100 x 10^9/L; Hb ≥ 90 g/L; serum Cr ≤ ULN; serum bilirubin ≤ 1.5 ULN; ALT/AST ≤ 1.5 ULN
6. Subjects should sign for the informed consent
7. Subjects should perform good compliance
8. Male and female subjects who have the ability of fertility should take contraception during the whole course and also 3 months after last dosage.In 7 days before the inclusion, urine pregnancy tests of subjects should be negative.

Exclusion Criteria:

1. Patients who have or are currently undergoing additional chemotherapy, radiation therapy or targeted therapy
2. Complete obstruction of the esophagus, or patients who have the potential to develop perforation
3. Patients with a history of malignancy (except that skin carcinomas or in situ breast cancer, oral cancer and cervical cancer with expected survival ≥2 years
4. Patients who multiple foci esophagus
5. Patients who are/were given any other medicine tests currently/in last 4 weeks
6. Experienced hypersensitiveness with similar medicine or other kinds of bio-medicines
7. Women in status of pregnancy
8. Patients who have complications exist as following:

(1)Uncontrolled angina and heart failure, have a history of hospitalization in 3 months; (2)A history of myocardial infarction in the past 6 months; (3)There is a need for antibiotic treatment of acute bacterial or fungal infection; (4)Chronic obstructive pulmonary disease, or other lung disease requiring hospitalization; (5)Drug addiction, alcoholism and AIDS disease or long-term virus carriers; (6)Uncontrollable seizures, or loss of insight because of mental illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2008-05; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | five years after enrollment
  failure: death from any cause

SECONDARY OUTCOMES:
Progression-free survival | five years after enrollment
  Failure: occurrence of local or regional progression, distant metastases, or death from any cause
local-regional control rate | three years after enrollment
  Failure: occurrence of local or regional progression
Adverse events | five years after enrollment
  assessed by RTOG Acute Radiation Morbidity Scoring Criteria and RTOG/EORTC Late Radiation Morbidity Scoring Schema
Health-related quality of life | five years after enrollment
  assessed by the Functional Assessment of Cancer Therapy-Esophageal (FACT-E)

CONTACTS AND LOCATIONS:
Overall Officials: Shixiu Wu, MD, Principal Investigator — 1st affliated hospital of Wen Zhou Medical college
Locations (1):
- 1st affliated hospital of Wen Zhou Medical college, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Xie C, Jing Z, Luo H, Jiang W, Ma L, Hu W, Zheng A, Li D, Ding L, Zhang H, Xie C, Lian X, Du D, Chen M, Bian X, Tan B, Xia B, Xie R, Liu Q, Wang L, Wu S. Chemoradiotherapy with extended nodal irradiation and/or erlotinib in locally advanced oesophageal squamous cell cancer: long-term update of a randomised phase 3 trial. Br J Cancer. 2020 Nov;123(11):1616-1624. doi: 10.1038/s41416-020-01054-6. Epub 2020 Sep 22. PMID 32958820